CLINICAL TRIAL: NCT05519969
Title: A Multicentre Audit of the Incidence of Pulmonary Aspiration With Different Fasting Regimens - European Preoperative Fasting Audit (EUROFAST)
Brief Title: A Multicentre Preoperative Fasting Audit
Acronym: EUROFAST
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Peter Frykholm, Assoc. Prof., Uppsala University
Other Study IDs: EUROFAST
Record Dates: First submitted 2022-08-22; First posted 2022-08-29 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Pulmonary Aspiration of Gastric Contents
Keywords: Preoperation fasting; General anesthesia; Children; Pulmonary aspiration of gastric contents
MeSH Terms: conditions — Respiratory Aspiration of Gastric Contents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 6-4-2 group: - Cases from centres implementing the rule of a minimum of 6 hours of fasting for solids, 4 hours for breast milk and 2 hours for clear fluids before anesthesia.
- 6-4-1 group: - Cases from centres implementing the 1 hour fasting rule for clear fluids recommended by ESAIC and specified in the guideline Preoperative fasting in children
- 6-4-0 group: - Cases from centres implementing the "zero" hour clear fasting rule, which means that children are allowed intake of clear fluids until they are called to the operating room

SUMMARY:
The new European Society of Anaesthesiology and Intensive Care (ESAIC) preoperative fasting guideline recommends a one hour minimum fasting time for clear fluids. This represents a major change in the practice of pediatric anaesthesia.

During the transition to shorter fasting times on a global scale, we need a large multicenter audit to monitor the incidence of pulmonary aspiration.

DETAILED DESCRIPTION:
The purpose of preoperative fasting is to achieve an empty stomach at the time of anaesthesia induction.

Most current fasting guidelines all take into account the balance between the risk of pulmonary aspiration and the harmful effects of prolonged preoperative fasting. However, there is increased awareness among pediatric as well as general anaesthesiologists that many patients suffer from prolonged duration of fasting in spite of the reasonable nominal respective limits of 6-4-2 hours. Prolonged fasting may be harmful, especially in small children, but also in adults with a poor nutritional status.

The new European Society of Anaesthesiology and Intensive Care (ESAIC, 2022) preoperative fasting guideline recommends a one-hour minimum fasting time for clear fluids. This represents a major change in the practice of paediatric anaesthesia. During the transition to shorter fasting times on a global scale, we need a large multicentre audit to monitor the incidence of pulmonary aspiration.

The primary aim of the European Preoperative Fasting Audit (EUROFAST) is to determine the safety of reducing the required fasting time for clear fluids to at least one hour in children fasting before elective procedures requiring general anaesthesia (as recommended in the ESAIC guideline).

ELIGIBILITY:
Inclusion Criteria:

* Children, age < 16 years old
* General anesthesia

Exclusion criteria

* Age > 15 years
* Procedure without general anesthesia
* General anesthesia performed at center with less than 1000 pediatric cases per year

Ages: 0 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children less than 16 years old
Sampling Method: Probability Sample
Enrollment: 307162 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Pulmonary aspiration | Intraoperative
  The incidence of confirmed pulmonary aspiration according to the study protocol

SECONDARY OUTCOMES:
Suspected pulmonary aspiration | Intraoperative
  The incidence regurgitation leading to transient desaturation that has resolved at the end of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Peter Frykholm, MD, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Plan to share data on request.
Supporting Information: Study Protocol
Time Frame: From ethics approval to Dec. 31, 2023
Access Criteria: Official web page
URL: https://www.uu.se/institution/kirurgiska-vetenskaper/forskning/anestesiologi-och-intensivvard/barnanestesi-och-perioperativ-medicin/eurofast

REFERENCES:
- See also: Pre-operative fasting in children: guideline from the European Society of Anaesthesiology and Intensive Care. — https://pubmed.ncbi.nlm.nih.gov/34857683/
- See also: Low incidence of pulmonary aspiration in children allowed intake of clear fluids until called to the operating suite — https://pubmed.ncbi.nlm.nih.gov/25940831/
- See also: Impact of clear fluid fasting on pulmonary aspiration in children undergoing general anesthesia: Results of the German prospective multicenter observational (NiKs) study — https://pubmed.ncbi.nlm.nih.gov/32533888/
- See also: Using quality improvement methods to reduce clear fluid fasting times in children on a preoperative ward — https://pubmed.ncbi.nlm.nih.gov/28675597/